CLINICAL TRIAL: NCT03976505
Title: Study of Comprehension and Execution of Medication Prescriptions Displayed on Touch-screens and Tablets in Parkinsonian Patients and Healthy Volunteers
Brief Title: Study of Comprehension and Execution of Medication Prescriptions in Parkinsonian Patients and Healthy Volunteers
Acronym: TACTIPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2017_843_0025
Record Dates: First submitted 2018-04-18; First posted 2019-06-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: medication prescriptions; eye-tracking; non-adherence; medication schedule
MeSH Terms: conditions — Parkinson Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: This study is exploratory, cross-sectional, experimental and monocentric. The experimental design is a split-plot 2(Group: parkinsonian patients vs. healthy volunteers) X 2(Condition: tablet vs. touch-screen + eye-tracker) X 2(Medication type: regular vs. irregular) X 2(Prescription format: table vs. textual) split-plot design in which Group and Condition are between-participants variables and Medication type and Prescription format are within-participants variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- textual prescription healthy volunteers (Active Comparator)
  Interventions: Other: reading a textual format prescription on a touch screen; Other: filling a virtual pillbox displayed on the screen as prescribed in the prescription; Other: eye-tracker; Other: cognitive tests and questionary
- table prescription healthy volunteers (Active Comparator)
  Interventions: Other: reading a table format prescription on a touch screen; Other: filling a virtual pillbox displayed on the screen as prescribed in the prescription; Other: eye-tracker; Other: cognitive tests and questionary
- textual prescription Parkinson's disease patients (Experimental)
  Interventions: Other: reading a textual format prescription on a touch screen; Other: filling a virtual pillbox displayed on the screen as prescribed in the prescription; Other: eye-tracker; Other: cognitive tests and questionary
- table prescription Parkinson's disease patient (Experimental)
  Interventions: Other: reading a table format prescription on a touch screen; Other: filling a virtual pillbox displayed on the screen as prescribed in the prescription; Other: eye-tracker; Other: cognitive tests and questionary

INTERVENTIONS:
Other: reading a table format prescription on a touch screen — Task consists in reading on a touch screen, or on a tablet, two fictive medication prescriptions. One is presented in a table format and the other in a textual format. Each prescription comprises two regular medications (same doses and moments of the day) and two irregular medications (different doses or different moments).
  Arms: table prescription Parkinson's disease patient; table prescription healthy volunteers
Other: reading a textual format prescription on a touch screen — Task consists in reading on a touch screen, or on a tablet, two fictive medication prescriptions. One is presented in a table format and the other in a textual format. Each prescription comprises two regular medications (same doses and moments of the day) and two irregular medications (different doses or different moments).
  Arms: textual prescription Parkinson's disease patients; textual prescription healthy volunteers
Other: filling a virtual pillbox displayed on the screen as prescribed in the prescription — filling a virtual pillbox displayed on the screen as prescribed in the prescription
Other: eye-tracker — In the touch-screen condition an eye-tracker is used to record eye fixations and scanpaths in real time.
Other: cognitive tests and questionary — Once the 2nd pillbox filling is finished a battery of cognitive tests and questionnaires is administered to participants to identify Pd subtypes of impaired performances.

SUMMARY:
Many patients with Parkinson's disease (Pd) don't respect medication prescriptions. Non-adherence is caused by several factors among which three play an important role: treatment complexity, cognitive decline, and patient-provider communication. One way for improving medication adherence in these patients is to identify the best way for adapting medication prescription presentation to these patients. This study is focused on prescriptions displayed on touch-screens and tablets.

This exploratory study aims at identifying the best format for presenting medication prescription to Pd patients. An experiment with Pd patients and healthy volunteers is carried out to analyze their behavior while filling a virtual pillbox from a education prescription presented electronically in different formats on a tablet or a touchscreen. A table format and a verbal format are compared to determine the most effective design for presenting medication schedules. A facilitating effect of the table format is hypothesized.

DETAILED DESCRIPTION:
Many Pd patients are non-adherent to their treatments. Because Pd patients are generally over 60 years old, suffer from cognitive disorders, and have complex medication regimens, taking medications as prescribed is a too complex cognitive task for them. It supposes the ability to understand the prescription, to plan and memorize the actions to carry out and to remember them while executing them. As prescriptions are communicated to patients via procedural documents, it should be possible to improve patient's comprehension by using a format suitable for their needs and characteristics. Previous studies with elderly people suggest that the table format is more effective than the textual format. However no study addressed this question with Pd patients.

One-hundred and twenty patients with Parkinson's disease and 120 healthy volunteers participate voluntarily to the study. Their task consists in reading on a touch screen, or on a tablet, two fictive medication prescriptions. One is presented in a table format and the other in a textual format. Each prescription comprises two regular medications (same doses and moments of the day) and two irregular medications (different doses or different moments). For each prescription, participants must fill a virtual pillbox displayed on the screen as prescribed in the prescription. Prescriptions and pillboxes are displayed by a tablet software specifically designed to record in real time all participant's actions and related chronometric data. Half participants perform the task in the " tablet condition ", and the other half in the " touch-screen " condition. In the touch-screen condition an eye-tracker is used to record eye fixations and scanpaths in real time. Once the 2nd pillbox filling is finished a battery of cognitive tests and questionnaires is administered to participants to identify Pd subtypes of impaired performances.

The main hypothesis predicts an effect of the format of prescriptions. More precisely, it consists in two concurrent hypotheses. H1a (the mental model model hypothesis): the table format should facilitate the pillboxes filling in the parkinsonian group and in the healthy volunteer group by facilitating the elaboration of an accurate mental model. H1b (the working memory load hypothesis): because parkinsonian patients are frequently impaired in visuospatial tasks, the tabular format could have no effect or could have a negative effect only in this group. A correlation between cognitive subtypes identified by cluster analyses and task performances is expected. Several secondary hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* all participants must have French as mother tongue,
* be able to sign the written informed consent form and must have reached the age of majority.
* Patients with Pd must have been diagnosed by a neurologist of the Amiens CHU (University Hospital Centre) more than 3 years ago, and must be in a ON period when participating to the two sessions.

Exclusion Criteria:

* photosensitive epilepsy,
* dyschromatopsias,
* not corrected visual acuity,
* dementia indicated by a Mini Mental State Examination score < 24,
* alcoholism or other drug addictions conditions known to impair mental status
* acute psychiatric or neurologic illness,
* failing to the training phase.
* Patients with Pd must not have other parkinsonian syndrome nor neurological, psychiatric or motor disorders, other than due to Pd.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Execution performance | 3 month
  concordance rate between prescription and pillbox filling

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No